CLINICAL TRIAL: NCT06158204
Title: A Randomized Controlled Crossover Lifestyle Intervention to Improve Metabolic & Mental Health in Female Healthcare Night Shift Workers
Brief Title: Improving Metabolic & Mental Health in Female Healthcare Shift Workers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Andrew Fruge, Associate Professor, Auburn University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 23-496 MR 2310
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-07

CONDITIONS: Sleep, Inadequate; Overweight and Obesity; Work Related Stress; Healthy Lifestyle
Keywords: circadian rhythm; protein; shift work; female; sleep
MeSH Terms: conditions — Sleep Deprivation; Overweight; Obesity; Occupational Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate intervention (Experimental): Participants will receive the 8-week intervention first, followed by 8 weeks of observation-only
  Interventions: Behavioral: Lifestyle Intervention
- Delayed intervention (Active Comparator): Participants will receive the 8-week intervention after 8 weeks of observation-only
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Behavioral: Lifestyle Intervention — Participants will receive guidance on when and what to eat and when to sleep and be physically active. Additionally, participants will be provided with whey protein isolate powder to be mixed with water and grain-based snack bars to be consumed primarily during work shifts. Lean body mass (kg) will be used to prescribe total caloric (~30kcal/kg lean mass) and protein (2g/kg lean mass) needs and sleep/rest goals will be 6-8 hours per 24 hour "day"

SUMMARY:
Circadian rhythm disruption caused by shift work alters metabolic and hormonal pathways, which accelerates chronic disease onset, leading to decreased quality and quantity of life. Preclinical studies indicate that optimizing nutrient and sleep/rest timing can mitigate these effects.

Female nightshift healthcare workers will be recruited to participate in a randomized crossover trial in which participants will be expected to follow the prescribed lifestyle intervention for eight weeks during the first or second eight-week periods of the study.

DETAILED DESCRIPTION:
Clinical assessments will include DEXA, phlebotomy, questionnaires, and stool collection, which will be completed at weeks 0, 8, and 16 to assess changes in metabolic health and quality of life. Four days of 24-hour dietary recalls will be collected at baseline, and weeks 4, 8, 12, and 16. Garmin Vivofit4 activity trackers will be provided to all participants at baseline, and participants will be reminded to sync the devices once weekly at minimum.

During the 8-week intervention phase, participants will receive guidance on when and what to eat and when to sleep and be physically active. Additionally, participants will be provided with whey protein isolate powder and grain-based snack bars to be consumed primarily during work shifts. Lean body mass (kg) will be used to prescribe total caloric (~30kcal/kg lean mass) and protein (2g/kg lean mass) needs and sleep/rest goals will be 6-8 hours per 24 hour "day."

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-50 years old
* BMI between 27 and 40 kg/m2
* >6 months in current predominantly night shift (average 30+ hours/week) schedule
* Can read and speak English
* Willing to correspond with study staff using smartphone technologies

Exclusion Criteria:

* Pregnant or undergoing hormonal treatment for fertility
* Major changes in any prescription medications within 3 months
* Major surgeries in last 3 months
* Diagnosis of Type 2 Diabetes or other major endocrine diseases
* Diagnosed food allergies or significant dietary limitations
* Currently engaged in intensive weight loss program
* Minimal medically necessary radiation exposure within the last year

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Visceral fat percentage | Change from 0-8 weeks; 8-16 weeks
  Change in visceral fat as a percentage of total fat mass as measured by dual x-ray absorptiometry. Lower values are optimal.
Mental Quality of Life | Change from 0-8 weeks; 8-16 weeks
  Research ANd Development (RAND) Short Form-12 will assess mental quality of life (Range 0-100; 100 is optimal).
Physical Quality of Life | Change from 0-8 weeks; 8-16 weeks
  Research ANd Development (RAND) Short Form-12 will assess physical quality of life (Range 0-100; 100 is optimal).

SECONDARY OUTCOMES:
Fasting serum triglycerides | Change from 0-8 weeks; 8-16 weeks
  Phlebotomy will be obtained while fasted 8+ hours and triglycerides will be measured as part of a comprehensive metabolic panel and reported in mg/dl. Lower concentrations are optimal.
Fasting alanine aminotransferase (ALT) | Change from 0-8 weeks; 8-16 weeks
  Phlebotomy will be obtained while fasted 8+ hours and alanine aminotransferase (ALT) will be measured as part of a comprehensive metabolic panel and reported in mg/dl. Lower concentrations are optimal.
Fasting serum blood glucose | Change from 0-8 weeks; 8-16 weeks
  Phlebotomy will be obtained while fasted 8+ hours and blood glucose will be measured as part of a comprehensive metabolic panel and reported in mg/dl. Lower concentrations are optimal.
Fasting serum low-density lipoproteins (LDL) | Change from 0-8 weeks; 8-16 weeks
  Phlebotomy will be obtained while fasted 8+ hours and low-density lipoproteins (LDL) will be measured as part of a comprehensive metabolic panel and reported in mg/dl. Lower concentrations are optimal.
Sleep - accelerometry | Change from 0-8 weeks; 8-16 weeks
  Average minutes of total daily sleep.
Total caloric intake | Change from 0-8 weeks; 8-16 weeks
  Four 24-hour dietary recalls will be obtained every four weeks and entered into the and analyzed in the Nutrition Data System for Research (NDSR).
Total protein intake | Change from 0-8 weeks; 8-16 weeks
  Four 24-hour dietary recalls will be obtained every four weeks and entered into the and analyzed in the Nutrition Data System for Research (NDSR).
Stool microbiome composition | Change from 0-8 weeks; 8-16 weeks
  16S changes in microbiome alpha diversity.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Frugé, PhD, Principal Investigator — Auburn University
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robinson LA, Lennon S, Pegel AR, Strickland KP, Feeley CA, Watts SO, J Van Der Pol W, Roberts MD, Greene MW, Fruge AD. A Randomized Controlled Crossover Lifestyle Intervention to Improve Metabolic and Mental Health in Female Healthcare Night-Shift Workers. Nutrients. 2025 Oct 24;17(21):3342. doi: 10.3390/nu17213342. PMID 41228416